CLINICAL TRIAL: NCT02002468
Title: Follow-up of Abnormal and Inadequate Test Results in the Danish Cervical Cancer Screening Program.
Brief Title: Follow-up of Abnormal and Inadequate Smear-test Results
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Cervix cancer screening
Record Dates: First submitted 2013-11-29; First posted 2013-12-05 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2015-12

CONDITIONS: Carcinoma in Situ of Uterine Cervix
Keywords: Risk Communication; Follow-up; Organisation of screening
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test result sent by letter (Experimental): The pap-smear test result is sent by letter directly to the women. Women in need of follow up are in the letter recommended to contact their general practitioner.
  Interventions: Other: Test result sent by letter; Other: Test result conveyed by general practitioners
- Test result conveyed by general practitioners (Active Comparator): In Denmark it is a standard procedure that general practitioners convey the pap-smear test results to the women.
  Interventions: Other: Test result conveyed by general practitioners

INTERVENTIONS:
Other: Test result sent by letter
  Arms: Test result sent by letter
Other: Test result conveyed by general practitioners

SUMMARY:
Denmark has a higher incidence of cervical cancer than other Nordic countries, although all Danish women (aged 23-65) are screened regularly to identify possible cervical dysplasia or asymptomatic invasive cancer.

Annually 40 000 women receives an abnormal or inadequate test result and a follow-up recommendation.

However problems with delayed follow-up may threaten the effectiveness of the Danish Cervical Cancer Screening Program, as 20% of women are delayed and dysplasia potentially can progress into cancer.

Delayed follow-up is found in situations where women either consciously or unconsciously postpone follow-up, or because of organizational aspects of the screening program, where communication regarding test results can fail either in content or with delay.This study will evaluate two interventions designed to increase follow-up:

1. A letter with the test result and potential recommendation for follow up will be sent to the women (RCT). The intention is to ensure that all women will be notified about the test result, quickly, homogenously and in layman's written language, still with the opportunity to contact or be contacted by the general practitioner, if there is special needs. Furthermore, it is assumed that general practitioner consultations regarding delivery of normal test results will decrease, so that cost savings is a potential side benefit
2. Electronic reminder to the general practitioner if women have not had the recommended follow up, giving the general practioner´s an opportunity to remind the women (retro perspective cohort study).

The results will be of great importance to the future organisation of cervical and colorectal cancer screening programmes in Denmark, but will also have international interest because of their similar challenges.

ELIGIBILITY:
Inclusion Criteria:

* woman with a pap-smear test

Exclusion Criteria:

* less than 23 years

Min Age: 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125000 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-10 (Actual); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of women with timely follow-up | 1½ year
  The proportion of women followed up will be calculated as cumulated incidence proportions according to four timeframes (undesirable early, as recommended, late, very late), and be compared by relative risks. The results will be presented in totals and separately depending on the test result (normal/inadequate/Bethesda classification 2001/HPV).

SECONDARY OUTCOMES:
Frequency of general practitioner contacts (consultations/telephone calls /e-mails) regarding conveying the smear test result. | Three months after the smear test.
  The two randomisation groups will be compared with respect to contacts with general practitioner after the smear test the first days, weeks, months after the general practitioner is notified of the screening result.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vedsted, Study Director — Center for Research in Cancer Diagnosis in Primary Care - (CaP), Aarhus University; Flemming Bro, Study Director — The Research Unit of General Practice in Aarhus, Aarhus University; Berit S Andersen, Study Director — The Department of Public Health Programmes at Regional Hospital Randers
Locations (1):
- University of Aarhus, Aarhus, Central Jutland, Denmark

REFERENCES:
- [Derived] Kristiansen BK, Andersen B, Bro F, Svanholm H, Vedsted P. Direct notification of cervical cytology results to women improves follow-up in cervical cancer screening - A cluster-randomised trial. Prev Med Rep. 2018 Nov 23;13:118-125. doi: 10.1016/j.pmedr.2018.11.015. eCollection 2019 Mar. PMID 30568870